CLINICAL TRIAL: NCT02050490
Title: Effect of the Implementation of a Symptom Diary on the Symptom Care Received and the Symptom Burden Experienced by Adult Cancer Patients Treated With Chemotherapy: A Before-and-after-study
Brief Title: Effect of a Symptom Diary on Symptom Care and Symptom Burden in Patients Treated With Chemotherapy: a Before-and-after-study
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other); Flemish League Against Cancer (Other); Onze Lieve Vrouw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B322201419701
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2016-10

CONDITIONS: Nausea; Vomiting; Pain; Anorexia; Etcetera
MeSH Terms: conditions — Nausea; Vomiting; Pain; Anorexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before group, no diary
- After group, with symptom diary

SUMMARY:
This study investigates whether the implementation of a symptom diary for reporting and communicating chemotherapy-related symptoms improves symptom care and decreases symptom burden in adult patients treated with chemotherapy.

The hypothesis is studied using a before-and-after design. First, symptom care and symptom burden will be observed in a sample of patients not being offered a symptom diary. Next, the symptom diary will be implemented at the participating hospital and symptom care and symptom burden will now be observed in a new sample of chemotherapy patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18) patients with (any type of) cancer treated with chemotherapy
* Understanding Dutch
* Being able to sign Informed consent

Exclusion Criteria:

* More than 3 lines of chemotherapy treatment in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18) patients with (any type of) cancer treated with chemotherapy
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
symptom distress | T1 (cycle 1, day 1), T2 (cycle 2, day 1), T3 (cycle 3, day 1), T4 (cycle 5, day 1)
  for each of 9 symptoms: how distressing was the symptom perceived by the patient? (ordinal variable)

SECONDARY OUTCOMES:
symptom severity | T1 (cycle 1, day 1), T2 (cycle 2, day 1), T3 (cycle 3, day 1), T4 (cycle 5, day 1)
  for each of 9 symptoms: how severe was the symptom? (ordinal variable)

OTHER OUTCOMES:
symptom care | T1 (cycle 1, day 1), T2 (cycle 2, day 1), T3 (cycle 3, day 1)
  binary variable expressing whether the patient has received care (either medication or advice) to help with the symptom

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Maria Middelares, Ghent, Belgium